CLINICAL TRIAL: NCT06967597
Title: Conservative Versus Proactive Management of Acute Cholecystitis After EUS-guided Transmural Gallbladder Drainage. Multicenter Randomized Clinical Trial: FUGITIVE Trial (FUGITIVE)
Brief Title: Conservative Versus Proactive Management of Acute Cholecystitis After EUS-guided Transmural Gallbladder Drainage: FUGITIVE Trial (FUGITIVE)
Acronym: FUGITIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General Universitario de Alicante (Other)
Responsible Party: Principal Investigator, Jose Ramon Aparicio Tormo, MD, Hospital General Universitario de Alicante
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CEIm Ref: 2024/141 (2024-0434)
Record Dates: First submitted 2025-05-03; First posted 2025-05-13 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Acute Cholecystitis
Keywords: EUS-guided gallbladder drainage; acute cholecystitis; interventional endoscopic ultrasonography; lumen apposing metal stents; percutaneous cholecystostomy
MeSH Terms: conditions — Cholecystitis, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cholecystoscopy, gallbladder cleaning and removal of lumen-apposing metal stent (Active Comparator): Elective upper gastrointestinal endoscopy to perform cholecystoscopy, cleaning and removal of gallbladder (GB) stones and retrieval of the Lumen Apposing Metal Stent (LAMS) will be conducted 1 month after endoscopic ultrasound-guided GB drainage. For persistent GB stones, consecutive procedures will be performed weekly until complete cleaning and retrieval of the LAMS. A coaxial double pigtail plastic stent (7 or 10 Fr x 3 cm) will be placed indefinitely to maintain the fistula between the GB and the digestive tract.
  Interventions: Procedure: Cholecystoscopy and gallbladder cleaning
- Conservative treatment: Indwelling stent (No Intervention): Patients in the conservative group will not be scheduled for endoscopic revision during the one-year follow-up. The LAMS will only be reviewed as part of routine practice for suspected LAMS related complications

INTERVENTIONS:
Procedure: Cholecystoscopy and gallbladder cleaning — Upper gastrointestinal endoscopy and cholecystoscopy are performed 4 weeks after GB drainage. A standard gastroscope is used to inspect the gallbladder cavity with retrieval or lithotripsy of residual stones until complete cleaning of the GB is achieved. Several procedures may be required to achieve complete stone clearance.
  Finally, the LAMS is retrieved and replaced with a double pigtail plastic stent.
  Arms: Cholecystoscopy, gallbladder cleaning and removal of lumen-apposing metal stent

SUMMARY:
Patients with gallbladder inflammation (acute cholecystitis) who cannot undergo surgery due to their fragility and surgical risk require a gallbladder drainage. It has been confirmed in previous studies that the gallbladder drainage from the digestive tract is a better alternative, because it has fewer complications than external (percutaneous) gallbladder drainage. However, there are no known studies that demonstrate whether it is better to maintain this drainage indefinitely, or to carry out periodic revisions of the drainage to progressively remove the stones lodged in the gallbladder and remove the drainage once this has been achieved. In this study we aim to compare the clinical evolution of patients who undergo this gallbladder drainage, dividing them into two groups:

* One group of patients in whom we maintain a metallic prosthesis or stent, which communicates the gallbladder with the stomach, indefinitely in order to always guarantee a drainage of the bile towards the digestive tract, and thus avoid new episodes of cholecystitis.
* Another group of patients who, one month after having undergone drainage, undergo a new procedure to remove the gallbladder lithiasis, until it is empty and without inflammation and we can remove the metal stent, leaving only a very thin plastic catheter to maintain the fistula and thus the bile continues to flow into the digestive tract. More than one procedure may be required to completely clear the gallbladder.

Knowledge of whether one strategy or the other presents fewer complications in the short, medium and long term is essential to be able to offer the best alternative to our patients.

The aim of the study is to compare the clinical outcome of these patients who have a definitive drain inserted with those who undergo several procedures to clear the gallbladder until the drain is removed. The rate of complications, the need for re-interventions and hospital admissions, new episodes of acute cholecystitis, quality of life and mortality of both groups over a period of one year are compared.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy is the gold standard for treating acute cholecystitis (AC). However, not all patients are suitable candidates for surgery during an AC episode. After recovery, some may improve sufficiently to undergo preventive surgery for future biliary events, while others remain high-risk surgical candidates or fail to recover adequately, making surgery infeasible. For these high-risk patients, optimal management remains uncertain. Currently, percutaneous drainage is the standard treatment, with endoscopic ultrasound-guided gallbladder drainage (EUS-GBD) emerging as a viable alternative in specialized centers. Recent data suggest that EUS-GBD may result in fewer complications compared to percutaneous drainage, with similar technical and clinical success rates.

Despite its promise, the optimal follow-up strategy for patients treated with EUS-GBD remains unclear, particularly regarding long-term complications associated with lumen-apposing metal stents (LAMS). Studies in pancreatic fluid collections suggest higher rates of complications, including bleeding and stent obstruction, leading to recommendations for early stent removal. However, for gallbladder drainage, the question arises whether LAMS should be maintained to prevent recurrence or replaced with less complication-prone stents like double pigtail stents.

The available evidence is contradictory. Some studies favor proactive endoscopic follow-up and gallstone removal to minimize recurrent cholecystitis, while others suggest that leaving LAMS indefinitely may reduce biliary events and hospital visits. To resolve these discrepancies, randomized prospective trials are needed to determine the optimal follow-up protocol for high-risk patients undergoing EUS-GBD for AC.

Our working hypothesis is that after EUS-GBD using a LAMS, there are no significant differences in the rate of biliopancreatic events between an active endoscopic approach (including gallbladder cleaning, stone extraction, and stent removal) and a conservative approach (without planned endoscopic interventions). Some studies even suggest that the proactive approach may lead to more complications The primary aim is to compare the rate of biliopancreatic events during one year of follow-up between patients treated with a proactive endoscopic strategy (group A) and those treated with a conservative strategy (group B) after EUS-GBD for acute cholecystitis (AC).

Secondary objectives focus on the evaluation of additional clinical outcomes, including complication rates at various time points, recurrence of biliary-related events, unplanned re-interventions, readmissions, mortality, disease-free survival, resolution of AC, and quality of life between the two groups.

This is a randomized, multicenter, open-label, nationwide, clinical trial. Patients will be randomized 1:1 to the two treatment groups stratified by center.

Centers eligible to participate as collaborating centers must have confirmed experience in EUS-guided procedures with EUS-GBD availability, having performed more than 10 EUS-GBD procedures prior to enrollment. Patient inclusion and exclusion criteria are specified in a separate section of the protocol.

For enrollment of patients, after diagnosis of AC, a patient evaluation by the surgical team or anesthesiologist declaring the patient unfit for surgery and the patient's willingness to undergo the EUS-GBD procedure is mandatory.

If the patient meets these requirements in addition to all previous inclusion criteria and none of the exclusion criteria, agrees to participate in the study, and signs the informed consent, the patient will be enrolled and randomized.

The randomization of patients to each of the treatment groups will be carried out centrally by the REDCap software; REDCap is a program that offers an online electronic data collection notebook. It will be stratified by center and by severity.

Patients will be randomized to two groups: Elective cholecystoscopy with stone extraction, eventual LAMS removal and double pigtail plastic stent (DPPS) placement or conservative management (indwelling LAMS). A total of 41 patients will be assigned to each group. In the group assigned to receive endoscopic interventions, upper gastrointestinal endoscopy will be programmed 4 weeks after de EUS-GBD and sequential procedures weekly thereafter until complete clearance of stones is achieved and the LAMS is removed and replaced with DPPS.

The procedure will be performed after at least 6 hours of fasting during the index admission, by endoscopists in charge of performing ERCP as usual in the collaborating centers under sedation controlled by endoscopists or anaesthesia according to the usual practice of the Endoscopy Unit of each collaborating center.

Gallbladder drainage will be performed with a LAMS, with a preference for stents ≥15 mm in diameter, and the preferred route will be duodenal (cholecystoduodenostomy); however, the final decision regarding stent size and route will be at the operator's discretion. After placement of the LAMS, a coaxial DPPS is placed. The DPPS complements the drainage and prevents complications.

After confirmation that the patient meets the inclusion criteria and none of the exclusion criteria, and after signing the informed consent form, the patient will undergo gallbladder drainage with a LAMS. The patient will then be randomized at their hospital to either group A (proactive treatment) or group B (conservative treatment). Randomization will not occur until after the drainage procedure has been completed.

Patient randomization in this clinical trial will be stratified by center to ensure an equal distribution of patients between the two intervention groups (proactive and conservative approaches) at each participating hospital. This stratification is essential to minimize potential center-specific differences that could influence outcomes.

Randomization sequences will be pre-generated using specialized software with blocks of four patients. Each block will randomly assign two patients to the proactive intervention group and two to the conservative group. This block design ensures that within each center, patients are sequentially and evenly assigned to both groups throughout the recruitment process, maintaining a constant balance. This approach is particularly critical because the trial may be stopped before the full expected sample size is reached.

The in-hospital management of patients with AC after EUS-GBD will be under the care of their attending physicians in the in-hospital ward of the respective collaborating center, who will follow the management recommended by the clinical guidelines. Their discharge will be decided by their regular physician. A clinical evaluation and laboratory tests will be performed 1 day and 7 days after the procedure (if the patient has not been discharged yet).

Periodic follow-up contacts are made: at 1 month, 6 months, 9 months, and 1 year. Contacts may be made by face-to-face or telematic visits after consultation with the patient, especially if the patient is institutionalized or has severe mobility problems. Additional laboratory tests are performed at the 1-month, 6-month and 1-year visits.

At these contacts, complications related to treatment and biliopancreatic events (BPE) that have occurred since the last visit are recorded. An interview will be conducted to record the presence of BPE that did not require admission (such as biliary colic or associated pain), recording the type and date of onset. The digital medical record will also be reviewed to record admissions and emergency department evaluations related or unrelated to BPE and to assess mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years of age
* Confirmed acute cholecystitis diagnosed according to Tokyo 2018 criteria.
* Patient unfit for surgery: if meets one or more of the following criteria: age ≥ 80 years, American Society of Anesthesiology (ASA) ≥ III, Charlson Comorbidity Index > 5 and/or Karnofsky < 50, or patient unwilling to undergo surgery.
* Gallbladder drainage by LAMS stent.
* Informed Consent signed

Exclusion Criteria:

* Patient refusal to participate in the study
* Gastrointestinal surgically modified anatomy preventing endoscopic access to the gallbladder.
* Technical failure to perform endoscopic ultrasound guided-gallbladder drainage.
* Moderate or severe ascites.
* Severe coagulopathy International Normalized Ratio >1.5 and/or fibrinogen <120) or thrombocytopenia (platelets <20,000).
* Patient unable to tolerate sedation or general anesthesia
* Haemodynamically unstable patient
* Life expectancy <6 months
* Baseline ECOG ≥4
* Patient with ongoing malignancy
* Pregnancy
* Acute pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Biliopancreatic events (BPE) | From enrollment until 12 months after
  The primary aim is to assess the difference in terms of recurrence of the combined variable of biliopancreatic events (biliary colic, cholangitis, choledocholithiasis, acute cholecystitis or acute pancreatitis) between the active treatment group and the conservative treatment group during follow-up period.

SECONDARY OUTCOMES:
Recurrence of each of the variables that make up the combined variable BPE separately | From enrollment until 12 months after
  To assess and compare the recurrence of each individual variable that constitutes the combined variable BPE across groups (AP, cholangitis, choledocholithiasis, cholecystitis, biliary colic)
Total complication rate | From enrollment until 12 months after
  The proportion of patients experiencing one or more complications during the study period
Unplanned reintervention rate | From enrollment until 12 months after
  The percentage of patients requiring unplanned additional surgical, radiologic or endoscopic interventions
Biliary cause admission rate | From enrollment until 12 months after
  The proportion of patients admitted to the hospital for biliary-related conditions
Disease-Free survival | From enrollment until 12 months after
  The time from treatment initiation to disease recurrence or death from any cause
Mortality rate | From enrollment until 12 months after
  The proportion of patients who die during the study period or within a defined follow-up time
Recurrence rate of cholecystitis | From enrollment until 12 months after
  The proportion of patients experiencing a new episode of cholecystitis after initial resolution
Clinical Success Rate for the Resolution of Cholecystitis | From enrollment until 12 months after
  The percentage of patients achieving complete resolution of cholecystitis symptoms with treatment

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Universitario Dr Balmis Alicante, Alicante, Alicante
  - Hospital General Universitario Dr. Balmis, Alicante, Alicante

IPD SHARING:
Plan to Share IPD: No